CLINICAL TRIAL: NCT00633880
Title: Phase III, Multi-Center, Study to Assess the Clinical Effect of Droxidopa in Subjects With Primary Autonomic Failure, Dopamine Beta Hydroxylase Deficiency or Non-Diabetic Neuropathy and Symptomatic NOH
Brief Title: Clinical Study of Droxidopa in Patients With Neurogenic Orthostatic Hypotension (NOH)
Acronym: NOH302
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chelsea Therapeutics (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Droxidopa NOH302
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-04

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypotension (NOH); Non-diabetic Neuropathy; Primary Autonomic Failure; Dopamine Beta Hydroxylase Deficiency
Keywords: NOH; Neurogenic Orthostatic Hypotension; Orthostatic hypotension; PAF; Pure Autonomic Failure; MSA; Multiple System Atrophy; Neuropathy; Autonomic Failure; Parkinson; Dopamine Deficiency; Dopamine; Droxidopa
MeSH Terms: conditions — dopamine beta hydroxylase deficiency; Hypotension, Orthostatic; Pure Autonomic Failure; Multiple System Atrophy | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Droxidopa (Experimental): Double-blind
  Interventions: Drug: Droxidopa
- Placebo (Placebo Comparator): Double-blind
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 100 mg, oral, three times per day 200 mg, oral, three times per day 300 mg, oral, three times per day 400 mg, oral, three times per day 500 mg, oral, three times per day 600 mg, oral, three times per day
  Arms: Placebo
Drug: Droxidopa — 100 mg, oral, three times per day 200 mg, oral, three times per day 300 mg, oral, three times per day 400 mg, oral, three times per day 500 mg, oral, three times per day 600 mg, oral, three times per day
  Other Names: L-DOPS; L-threo-DOPS; Northera
  Arms: Droxidopa

SUMMARY:
The purpose of this study is to see whether droxidopa is effective in treating symptoms of neurogenic orthostatic hypotension in patients with Primary Autonomic Failure (Pure Autonomic Failure, Multiple System Atrophy, Parkinson's Disease), Non-diabetic neuropathy, or Beta Hydroxylase deficiency.

DETAILED DESCRIPTION:
Systolic blood pressure is transiently and minimally decreased in healthy individuals upon standing. Normal physiologic feedback mechanisms work through neurally-mediated pathways to maintain the standing blood pressure, and thus maintain adequate cerebral perfusion. The compensatory mechanisms that regulate blood pressure upon standing are dysfunctional in subjects with orthostatic hypotension (OH), a condition that may lead to inadequate cerebral perfusion with accompanying symptoms of syncope, dizziness or lightheadedness, unsteadiness and blurred or impaired vision, among other symptoms.

The autonomic nervous system has a central role in the regulation of blood pressure. Primary Autonomic Failure is manifested in a variety of syndromes. Orthostatic hypotension is a usual presenting symptom. Primary Autonomic Failure may be the primary diagnosis, and classifications include pure autonomic failure (PAF), also called idiopathic orthostatic hypotension (Bradbury-Eggleston syndrome) autonomic failure with multiple system atrophy (Shy-Drager syndrome) and also Parkinson's disease. Regardless of the primary condition, autonomic dysfunction underlies orthostatic hypotension.

Orthostatic hypotension may be a severely disabling condition which can seriously interfere with the quality of life of afflicted subjects. Currently available therapeutic options provide some symptomatic relief in a subset of subjects, but are relatively ineffective and are often accompanied by severe side effects that limit their usefulness. Support garments (tight-fitting leotard) may prove useful in some subjects, but is difficult to don without family or nursing assistance, especially for older subjects. Midodrine, fludrocortisone, methylphenidate, ephedrine, indomethacin and dihydroergotamine are among some of the pharmacological interventions that have been used to treat orthostatic hypotension, although only midodrine is specifically approved for this indication. The limitations of these currently available therapeutic options, and the incapacitating nature and often progressive downhill course of disease, point to the need for an improved therapeutic alternative.

The current withdrawal design study will measure the efficacy of droxidopa on symptoms of neurogenic orthostatic hypotension in patients randomized to continued droxidopa treatment versus placebo, following 14 days of double-blind treatment.

droxidopa

droxidopa [also, known as L-threo-3,4-dihydroxyphenylserine, L-threo-DOPS, or L-DOPS] is the International non-proprietary name (INN) for a synthetic amino acid precursor of norepinephrine (NE), which was originally developed by Sumitomo Pharmaceuticals Co., Limited, Japan. It has been approved for use in Japan since 1989. Droxidopa has been shown to improve symptoms of orthostatic hypotension that result from a variety of conditions including Shy Drager syndrome (Multiple System Atrophy), Pure Autonomic Failure, and Parkinson's disease. There are four stereoisomers of DOPS; however, only the L-threo-enantiomer (droxidopa) is biologically active.

The exact mechanism of action of droxidopa in the treatment of symptomatic NOH has not been precisely defined; however, its NE replenishing properties with concomitant recovery of decreased noradrenergic activity are considered to be of major importance.

Droxidopa has been marketed in Japan since 1989. Data from clinical studies and post-marketing surveillance programs conducted in Japan show that the most commonly reported adverse drug reactions with droxidopa are increased blood pressure, nausea, and headache. In clinical studies, the prevalence and severity of droxidopa adverse effects appear to be similar to those reported by the placebo control arm.

ELIGIBILITY:
PATIENT INCLUSION CRITERIA:

* Male or female and aged 18 years or over;
* Clinical diagnosis of orthostatic hypotension associated with Primary Autonomic Failure (PD, MSA and PAF), Dopamine Beta Hydroxylase Deficiency or Non-Diabetic Autonomic Neuropathies;
* A documented fall in systolic blood pressure of at least 20 mmHg, or in diastolic blood pressure of at least 10 mmHg, within 3 minutes after standing;
* Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care.

MAIN PATIENT EXCLUSION CRITERIA:

* Taking ephedrine or midodrine; Patients taking ephedrine or midodrine may enroll after a minimum 7 day washout period;
* Taking anti-hypertensive medication;
* Have a history of more than moderate alcohol consumption;
* Women who are pregnant or lactating;
* Have a history of closed angle glaucoma;
* Have pre-existing sustained severe hypertension (BP > 180/110 mmHg in the sitting position);
* Have atrial fibrillation or, in the investigator's opinion, have any other significant cardiac arrhythmia;
* In the investigator's opinion, have any other significant systemic, hepatic, cardiac or renal illness;
* Have diabetes mellitus or insipidus;
* Have a known or suspected malignancy;
* Have known gastrointestinal illness or other gastrointestinal disorder that may, in the investigator's opinion, affect the absorption of study drug;
* In the investigator's opinion, have clinically significant abnormalities on clinical examination or laboratory testing;
* Have a serum creatinine level > 130 µmol/L;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, MD, Principal Investigator — NYU Langone Health; Christopher J Mathias, MD, Principal Investigator — Imperial School of Medicine; Roy Freeman, MD, Principal Investigator — Harvard Medicine School; Phillip A Low, MD, Principal Investigator — Mayo Foundation
Locations (54):
- United States (44):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Dedicated Clinical Research, Litchfield Park, Arizona
  - Xenoscience Inc., Phoenix, Arizona
  - Sun Health Research Institute, Sun City, Arizona
  - The Parkinson's and Movement Disorders Institute, Fountain Valley, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - The Parkinson's Institute, Sunnyvale, California
  - Electrophysiology Associates, Colorado Springs, Colorado
  - Parkinson's Disease & Movment Disorder Center, Boca Raton, Florida
  - Southeastern Integrated Medical, Gainesville, Florida
  - Mayo Jacksonville Florida Department of Neurology, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Medical Associates of North Georgia, Canton, Georgia
  - Saint Mary of Nazareth Hospital Center, Chicago, Illinois
  - North Chicago VA Medical Center, North Chicago, Illinois
  - Indiana Medical Research, Elkhart, Indiana
  - JWM Neurology, Indianapolis, Indiana
  - Kansas City Bone and Joint, PA, Overland Park, Kansas
  - University of Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Henry Ford Health System, Southfield, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - New Jersey Neuroscience Institute, Edison, New Jersey
  - Kingston Neurological Associates, PC, Kingston, New York
  - NYU Medical Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - Jacinto Medical Group, PA, Baytown, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Scott & White Healthcare - Round Rock, Round Rock, Texas
  - Scott & White Memorial Hospital & Clinic, Temple, Texas
  - East Texas Medical Center, Tyler, Texas
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Baker Heart Research Institute, Melbourne, Victoria
  - Austin Hospital, Heidelburg
- Canada (5):
  - McMaster University, Hamilton, Ontario
  - Centre for Movement Disorders, Markham, Ontario
  - Parkinson's & Neurodegenerative Disorders Clinic, Ottawa, Ontario
  - SMBD Jewish General Hospital, Montreal, Quebec
  - Quebec Memory and Motor Skills Disorders Clinic, Québec, Quebec
- New Zealand (2):
  - Auckland Hospital, Grafton Auckland, Private Bag
  - Van der Veer Institute for Parkinson's Disease and Movement Disorders, Christchurch

REFERENCES:
- [Derived] Biaggioni I, Arthur Hewitt L, Rowse GJ, Kaufmann H. Integrated analysis of droxidopa trials for neurogenic orthostatic hypotension. BMC Neurol. 2017 May 12;17(1):90. doi: 10.1186/s12883-017-0867-5. PMID 28494751
- [Derived] Francois C, Rowse GJ, Hewitt LA, Vo P, Hauser RA. Analysis of number needed to treat for droxidopa in patients with symptomatic neurogenic orthostatic hypotension. BMC Neurol. 2016 Aug 18;16(1):143. doi: 10.1186/s12883-016-0665-5. PMID 27538531
- [Derived] Biaggioni I, Freeman R, Mathias CJ, Low P, Hewitt LA, Kaufmann H; Droxidopa 302 Investigators. Randomized withdrawal study of patients with symptomatic neurogenic orthostatic hypotension responsive to droxidopa. Hypertension. 2015 Jan;65(1):101-7. doi: 10.1161/HYPERTENSIONAHA.114.04035. Epub 2014 Oct 27. PMID 25350981

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Titration: All patients titrated to their optimal dose of droxidopa during an initial open label phase for 7-14 days
Period: Open Label Titration
Arm/Group | Open Label Titration | Droxidopa | Placebo
Started | 181 | 0 | 0
Completed | 101 | 0 | 0
Not Completed | 80 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Adverse Event | 13 | 0 | 0
Not completed — Treatment Failure | 55 | 0 | 0
Not completed — Protocol Violation | 6 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Period: Randomized Double Blind
Arm/Group | Open Label Titration | Droxidopa | Placebo
Started | 0 | 50 | 51
Completed | 0 | 50 | 51
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized: Entered open-label droxidopa dose titration, but did not randomize
- Total: Total of all reporting groups
Arm/Group | Not Randomized | Droxidopa | Placebo | Total
Number analyzed (Participants) | 80 | 50 | 51 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (9.74) | 63.1 (13.76) | 66.6 (11.25) | 66.9 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 20 | 19 | 74
  Male | 45 | 30 | 32 | 107
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 80 | 49 | 49 | 178
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 25 | 32 | 110
  Canada | 8 | 9 | 2 | 19
  United Kingdom | 5 | 3 | 2 | 10
  Poland | 5 | 10 | 8 | 23
  Australia | 8 | 2 | 6 | 16
  New Zealand | 1 | 1 | 1 | 3
Primary Clinical Diagnosis [Number; unit: participants]
  Parkinson's Disease | 38 | 21 | 23 | 82
  Multiple System Atrophy | 21 | 17 | 13 | 51
  Pure Autonomic Failure | 18 | 8 | 10 | 36
  Dopamine Beta-Hydroxylase Deficiency | 0 | 0 | 1 | 1
  Non-Diabetic Autonomic Neuropathy | 2 | 2 | 3 | 7
  Other | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Dizziness/ Lightheadedness/ Feeling Faint/ or Feeling Like You Might Blackout (OHSA Item 1)
Description: OHSA item 1 scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug) .
Time Frame: 14 days
Population: Missing data were imputed using the last observation carry forward method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 50 | 51
units on a scale | 1.3 (2.75) | 1.9 (3.16)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.509, Wilcoxon (Mann-Whitney) — Statistical analysis plan involved a hierarchical assessment of secondary endpoints to prevent inflation of type I errors. As the primary endpoint was not positive, statistical analysis was not performed on secondary endpoints

2. Secondary Outcome: Change in Fatigue (OHSA Item 4)
Description: OHSA item 4 scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug) .
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 50 | 51
units on a scale | 0.7 (2.61) | 1.5 (2.72)

3. Secondary Outcome: Change in Weakness (OHSA Item 3)
Description: OHSA item 3 scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug) .
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 50 | 51
units on a scale | 0.3 (2.88) | 1.2 (2.70)

4. Secondary Outcome: Change in Vision (OHSA Item 2)
Description: OHSA item 2 scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug) .
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 50 | 51
units on a scale | 1.1 (2.79) | 0.8 (2.24)

5. Secondary Outcome: Change in Concentration (OHSA Item 5)
Description: OHSA item 5 scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug) .
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 50 | 51
units on a scale | 0.1 (2.74) | 0.9 (2.67)

6. Post Hoc Outcome: Change in Orthostatic Hypotension Questionnaire Score (OHQ)
Description: The OHQ is the average of two sub-scales, the Orthostatic Hypotension Symptom Assessment Scale (OHSA) and the Orthostatic Hypotension Daily Activities Scale (OHDAS). Each asks the patient to rate their symptoms or disease impact over the past week. The OHSA sub-scale is the average of six items: 1) Dizziness, lightheadedness, feeling faint or feeling like you might black out; 2) Problems with vision; 3) Weakness; 4) Fatigue; 5) Trouble concentrating; and 6) Head/neck discomfort. The OHDAS sub-scale is the average of four items: 1) Standing for a short time; 2) Standing for a long time; 3) Walking for a short time; and 4) Walking for a long time. Each item is scored on a Likert scale from 0 to 10, with 10 being the most severe.
  In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug) .
Time Frame: 14 days
Population: 3 droxidopa patients and 2 placebo patients were excluded from the analysis due to missing randomization values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 47 | 49
units on a scale | 0.11 (2.176) | 1.22 (2.390)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.026, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Change in Head/Neck Discomfort (OHSA Item 6)
Description: OHSA item 6 scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug) .
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 50 | 51
units on a scale | -0.1 (2.45) | 1.2 (3.19)

8. Secondary Outcome: Change in Ability to Conduct Activities of Daily Living Score (OHDAS Composite Score)
Description: The OHDAS scale is the average of four items: 1) Standing for a short time; 2) Standing for a long time; 3) Walking for a short time; and 4) Walking for a long time. Each asks the patient to rate their disease impact over the past week. Each item is scored on a Likert scale from 0 to 10, with 10 being the most severe. Change: score at end of study minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug) .
Time Frame: 14 days
Population: One placebo patient excluded from analysis because OHDAS values were not evaluable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 50 | 50
units on a scale | -0.24 (2.35) | 0.91 (2.50)

9. Secondary Outcome: Change in Orthostatic Hypotension Symptom Assessment Score (OHSA Composite)
Description: The OHSA scale is the average of six items: 1) Dizziness, lightheadedness, feeling faint or feeling like you might black out; 2) Problems with vision; 3) Weakness; 4) Fatigue; 5) Trouble concentrating; and 6) Head/neck discomfort. Each asks the patient to rate their symptoms over the past week. Each item is scored on a Likert scale from 0 to 10, with 10 being the most severe. Change: score at end of study minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug) .
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 50 | 51
units on a scale | 0.6 (2.27) | 1.35 (2.53)

10. Secondary Outcome: Change in Orthostatic Hypotension Symptom Scores Excluding Dizziness (OHSA Composite Items 2-6)
Description: OHSA composite scale (items 2-6) is the average of five OHSA items: 2) Problems with vision; 3) Weakness; 4) Fatigue; 5) Trouble concentrating; and 6) Head/neck discomfort. Each asks the patient to rate their symptoms over the past week. Each item is scored on a Likert scale from 0 to 10, with 10 being the most severe. Change: score at end of study minus score at randomization. In this withdrawal design, a positive score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug) .
Time Frame: 14 days
Population: One placebo patient excluded from analysis per the SAP because all baseline values in the composite were zero.
  LOCF was used to impute values for patients who did not have an end of study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 50 | 50
units on a scale | 0.44 (2.29) | 1.07 (2.25)

11. Secondary Outcome: Change in Systolic Blood Pressure (SBP) Measurements 3 Minutes Post Standing;
Description: Change: standing systolic blood pressure at end of study minus standing systolic blood pressure at randomization. In this withdrawal design, a negative score indicates worsening during the double-blind randomized phase relative to value at randomization (on open-label drug) .
Time Frame: 14 days
Population: three placebo patients excluded from the analysis due to missing standing blood pressure values at either randomization or end of study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 50 | 48
mmHg | -7.6 (19.71) | -5.2 (26.83)

ADVERSE EVENTS:
Groups:
- Open Label Phase: All patient titrated on droxidopa during open-label phase
Arm/Group | Droxidopa | Placebo | Open Label Phase
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/51 | 4/181
Other Adverse Events (participants affected / at risk) | 4/50 | 11/51 | 44/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Droxidopa (N=50) | Placebo (N=51) | Open Label Phase (N=181)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Droxidopa (N=50) | Placebo (N=51) | Open Label Phase (N=181)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 20 (28)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 15 (18)
Fatigue (General disorders) | 0 (0) | 1 (1) | 10 (10)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 6 (7) | 9 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less